CLINICAL TRIAL: NCT03137524
Title: A Pilot Study of Hand-held Fan Therapy in Breathless Chronic Obstructive Pulmonary Disease (COPD) Patients
Brief Title: Fan Therapy in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 218706
Record Dates: First submitted 2017-04-24; First posted 2017-05-02 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Breathlessness
Keywords: Fan or Air Therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Intervention Model Description: Single Centre Pilot study using a randomised controlled crossover design (aka randomised A-B single-subject design).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Held Fan Therapy (Experimental)
  Interventions: Device: Hand Held Fan Therapy
- No Intervention (No Intervention)

INTERVENTIONS:
Device: Hand Held Fan Therapy — Hand-Held fan therapy used to generate airflow directed to face during specific exercise test
  Arms: Hand Held Fan Therapy

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common smoking related lung disease. The main symptom in breathlessness.

Pulmonary Rehabilitation (PR) - a supervised group exercise and education class - is an effective intervention in COPD to reduce symptoms, improve exercise performance and prevent exacerbations. However some COPD patients are unable to to effectively exercise as they are limited by their breathlessness, despite optimal medical management. By reducing their physical activity to avoid the onset of breathlessness, they become deconditioned and then further attempts at exercise make them more breathless, leading to an inactivity cycle.

There is a growing evidence base regarding the use of hand hold fan therapy or air therapy to relieve breathlessness at rest. Limited studies have looked at the use of fan therapy during exercise, and its role on exercise capacity and recovery time, provisional results which indicate it may also be useful during activity. Logically you might expect patients who are less breathless to be able to exercise more, or recover quicker.

This study aims to investigate the effects a hand held fan will have on sensation of breathlessness and exercise capacity in patients with COPD. This will involve participants undertaking a standardised field walking test ( 6 minute walk test) with and with out the fan and then comparing the distance covered and how they felt during and after exercise. This will better inform how we structure exercise and advice to these patients in the future to empower patients limited by breathlessness.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease (Forced Expiratory volume in 1 second (FEV1)/Vital capacity ratio < 70%, with an observed respiratory impairment ( Global initiative for Chronic Obstructive Lung Disease (GOLD) stage II-IV: < 79% FEV1 predicted)
* Age > 18 years old
* Exertional breathlessness with a Medical Research Council (MRC) breathlessness scale greater of equal to 2

Exclusion Criteria:

* Recent exacerbation of COPD symptoms requiring antibiotics within the preceding 4 weeks
* Significant cardiovascular or peripheral disease that could influence exercise tolerance and ability to perform exercise test
* Unable to hold fan to face and mobilise
* On Long Term Oxygen Therapy or fulfils criteria for ambulatory oxygen
* Lack of English Language Competency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-07-26 (Actual); Study Completion 2017-07-26 (Actual)

PRIMARY OUTCOMES:
Breathlessness as measured on the Numerical Rating Scale (NRS) | Change from baseline measurement of breathlessness on the NRS to the measurement of breathlessness on NRS after a 6 minute walk test
  Units on a Scale

SECONDARY OUTCOMES:
Walking distance | 6 minutes
  as measured during a 6 minute walk test
Oxygen Saturation Levels | 6 minutes
  peripheral oxygen saturation levels as measured during a 6 minute walk test
Recovery time | in minutes, anticipate no longer than 10minutes
  Time in mins taken for sensation of breathlessness to return to baseline levels after completion of a 6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dr Cartwright, BSc, MSc, PhD, Principal Investigator — City, University of London
Locations (1):
- King's College Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Long A, Cartwright M, Reilly CC. Impact of fan therapy during exercise on breathlessness and recovery time in patients with COPD: a pilot randomised controlled crossover trial. ERJ Open Res. 2021 Nov 8;7(4):00211-2021. doi: 10.1183/23120541.00211-2021. eCollection 2021 Oct. PMID 34760995